CLINICAL TRIAL: NCT07127614
Title: The Relationship Between Primary Tumor Depth of Invasion and Neck Lymph Nodes Management in T1T2N0 Oral Cavity Squamous Cell Carcinomas
Brief Title: Primary Tumor Depth of Invasion and Lymph Node Management in Oral Squamous Cell Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Islam Mohamed Mohamed Ali, Assistant Lecturer, Al-Azhar University
Other Study IDs: 1008/2042
Record Dates: First submitted 2025-07-30; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Squamous Cell Carcinoma Mouth
Keywords: squamous cell carcinoma; MRI; diagnostic accuracy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biopsy from the tumor will be retained as fixed tissues to undergo the histopathological examination and determination of the pathological depth of invasion

GROUPS / COHORTS (1):
- study group: Patients with biopsy proven oral squamous cell carcinoma with the edition T1or T2 N0 based on TNM staging by American Joint cancer center AJCC 8th edition
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Histo-Pathological examination of the resected tumor tissues

INTERVENTIONS:
Diagnostic Test: MRI — pre-operative MRI scan
  Other Names: index test
Diagnostic Test: Histo-Pathological examination of the resected tumor tissues — histo-pathological examination of the resected tumor tissues with the lymph nodes involved to determine the pathological depth of invasion
  Other Names: Reference test

SUMMARY:
To evaluate the diagnostic accuracy of preoperative MRI in the determination of the primary tumor depth of invasion (DOI) as a predictor factor in neck lymph nodes management in T1T2N0 oral cavity squamous cell carcinomas as compared to the pathological depth of invasion

DETAILED DESCRIPTION:
A diagnostic accuracy study comparing preoperative MRI scans to pathological examination of the resected oral squamous cell carcinoma with lymph nodes to determine the depth of invasion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven oral squamous cell carcinoma with the edition T1or T2 N0 based on TNM staging by the American Joint Cancer Center AJCC 8th edition
* The primary tumor has a depth of invasion (DOI) greater than 4 mm
* Clinical N0 status confirmed by reasonable parameters includes computed tomography CT, MRI, -Ultrasonography,( US fine needle aspiration in suspected lymph nodes )
* The primary tumor must be reliably resected to a clear margin without the need for entry of the neck for reconstruction

Exclusion Criteria:

* Patients with T3T4 OCSCC
* Proven or suspected positive neck node
* Patient with distant metastasis
* Patient with gross injury to the neck that precludes proper surgical dissection.
* Patient with a history of radiotherapy to the neck
* Recurrent cases of OCSCC or recurrent node disease
* Patient with previous neck node biopsy or previous neck dissection
* Patient with a medical condition or performance that interferes with the surgical intervention as judged by the specialist physician

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with biopsy-proven oral squamous cell carcinoma with the edition T1or T2 N0 based on TNM staging by the American Joint Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | immediately after the surgery
  determination of the diagnostic accuracy of MRI in determining the depth of invasion compared to the pathological depth of invasion

CONTACTS AND LOCATIONS:
Overall Officials: Wael A ElMohandes, PhD, Study Director — oral and maxillofacial surgery, Faculty of Dental Medicine, Al-Azhar University; Ahmed M Alfar, PhD, Study Chair — oral and maxillofacial surgery, Faculty of Dental Medicine, Al-Azhar University; Mohamed A Mohamed, PhD, Study Chair — oral and maxillofacial surgery, Faculty of Dental Medicine, Al-Azhar University; Mohamed AW Amin, PhD, Study Chair — oral and maxillofacial surgery, Faculty of Dental Medicine, Al-Azhar University
Locations (1):
- AL Sayed Galal Hospital Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Finished results will be published in a scientific journal
Supporting Information: Study Protocol
Time Frame: beginning after publication and for 6 months ending
Access Criteria: IPD data will be made available upon reasonable request from the principal investigator.